CLINICAL TRIAL: NCT00108173
Title: Neural Substrates of Treatment for Nicotine Dependence
Brief Title: Brain Reaction to Treatment of Nicotine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ADRD-018-02S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Nicotine Dependence
Keywords: Position Emission Tomography (PET); Nicotine dependence; functional magnetic resonance imaging; cigarette cues
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Zyban

INTERVENTIONS:
Drug: Zyban

SUMMARY:
The purpose of the study was to determine how the treatments for cigarette craving work.

Hypothesis: During exposure to cigarette-related cues, heavy smokers will have greater reductions in regional brain activation from before to after both forms of active treatments than from before to after placebo.

DETAILED DESCRIPTION:
PET and fMRI scanning were used to examine brain activity and activation in cigarette smokers in response to cigarette-related cues.

ELIGIBILITY:
Inclusion Criteria:

* Heavy smoker, more than one pack per day
* Free of medical conditions or medications that affect brain activity
* Not pregnant

Exclusion Criteria:

Drug or alcohol dependence Mental Illness Pregnancy Medications that affect brain function Unstable medical conditions

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2002-10; Primary Completion 2007-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
2-FA PET scan results | Within the first few weeks of study initiation
  Brain activity and activation in response to cigarette-related cues

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L. Brody, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States